CLINICAL TRIAL: NCT06214468
Title: Protective Effect of Nicotinamide Riboside Against Acetaminophen Toxicity
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Alabama (Other)
Collaborators: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency); University of Nevada, Las Vegas (Other); University of Alabama at Birmingham (Other); Rutgers University (Other)
Responsible Party: Principal Investigator, Marie Migaud, Professor of Pharmacology, University of South Alabama
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 23-067/2026659-2
Record Dates: First submitted 2023-12-07; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Drug Toxicity
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Acetaminophen; nicotinamide-beta-riboside; Niacinamide

STUDY DESIGN:
Intervention Model Description: This study takes place over 2 days, and the study runs twice, two weeks apart. Upon enrolment and consent, the participant will provide a urine sample then be given acetaminophen and Nicotinamide Riboside (NR). Participant are asked to collect 4 urine samples over a 24 hour period and record the time of the collection each time. Two weeks after this first collection, participants are asked to repeat the process but this time with only acetaminophen ingestion.
  Tubes will be provided for the collection of the urine and zip lock bags will be provided to place the tubes in after samples have been collected. All samples should be stored in the freezer until completion of the samples at which time they should be brought to the USA Mitchell Cancer Institute. Some volunteers will participate in 4 total blood draws collected on the first day at the time of the consent then again 6 hours after taking NR and Acetaminophen. Blood samples will be taken again during the second collection period.
Who Masked: Participant, Investigator
Masking Description: Sample will be assigned a unique identifier to de-identify samples from the study team. This unique identifier will be assigned by the clinical manager, who will be providing the informed consent. Each sample will be labeled to include gender, race and ethnicity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tylenol and Nicotinamide Riboside (Other)
  Interventions: Combination Product: Acetaminophen and Nicotinamide Riboside; Drug: Acetaminophen
- Tylenol Only (Active Comparator)
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Combination Product: Acetaminophen and Nicotinamide Riboside — Collection of urine at different time intervals following ingestion of Tylenol plus Nicotinamide Riboside
  Other Names: Tylenol and Vitamin B3
  Arms: Tylenol and Nicotinamide Riboside
Drug: Acetaminophen — Collection of urine at different time intervals following ingestion of Tylenol only
  Other Names: Tylenol

SUMMARY:
Over-the-counter drugs like acetaminophen (e.g., Tylenol®) can be detrimental. In space, astronauts who have pain and constant discomfort use acetaminophen extensively. Investigators are studying the effects of acetaminophen under space-like conditions since acetaminophen might affect astronauts' health. Investigators also wish to see whether a dietary supplement can reduce some negative effects of acetaminophen.

It is believed that acetaminophen promotes the productions of chemicals in the body that could be toxic.

In this study, measurements of these chemicals in urine after ingestion of 1 tablet of acetaminophen and compare these measurements to when acetaminophen is taken at the same time as a dietary supplement. This study will also explore whether these products are more abundant when blood is placed under conditions that mimic space. Therefore, this study will collect blood from a few volunteers who took acetaminophen, and acetaminophen with the dietary supplement.

DETAILED DESCRIPTION:
In space, astronauts are constantly exposed to conditions the body is not used to. To relieve pain and discomfort, astronauts often use acetaminophen. This study investigates a possible negative synergistic effect between using acetaminophen and space-like stressors as they both generate oxidative stress and produce toxins that distribute around the body and disrupt cellular function in other tissues. The study seeks to examine whether a dietary supplement, nicotinamide riboside (NR), can reduce some adverse effects of these toxins by reducing their production when taking acetaminophen.

The study will measure these materials in urine after ingestion of 1 gram of acetaminophen and compare these measurements to when the same amount of acetaminophen is taken at the same time as NR. It will also evaluate whether these toxins are more abundant when blood is placed under conditions resembling space. Therefore, blood collection from a few volunteers who take acetaminophen, and acetaminophen with NR. Ultimately, this work will establish whether NR could reduce the generation of specific endotoxins.

For this study, male and female volunteers are needed to donate urine for testing the effect of 1000mg dose of Tylenol® and one 1000mg dose of Tylenol® with one 250mg dose of Nicotinamide Riboside on the abundance of uremic toxins in urine and in blood. Volunteers are also needed to donate blood.

ELIGIBILITY:
Inclusion Criteria:

* n/a

Exclusion Criteria:

* Individual allergic to acetaminophen or nicotinamide riboside

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Count the quantity of NAD(P)(H) present with exposure to acetaminophen, with and without NR | At consent and 6 hours post dose
  Multiple blood draws pre and post dose of acetaminophen plus NR
Count the DNA damage occurring upon space-like stressors following exposure to acetaminophen, with and without NR | At consent and 6 hours post dose
  Multiple blood draws pre and post dose of acetaminophen with or without NR.
Count the quantity of ox-NAD(P) present with exposure to acetaminophen, with and without NR | At consent and 6 hours post dose
  Multiple blood draws pre and post dose of acetaminophen plus NR
Count the quantity of PYR-ribosides present with exposure to acetaminophen, with and without NR | Pre-dose and 6 hour, 12 hour and 24 hour post dose following administration and
  A urine sample will be collected from consented volunteers pre and post dose of acetaminophen plus NR
Count the quantity of PYR-nucleotides present with exposure to acetaminophen, with and without NR | Pre-dose and 6 hour, 12 hour and 24 hour post dose following administration and
  A blood sample will be collected from consented volunteers pre and post dose of acetaminophen plus NR

CONTACTS AND LOCATIONS:
Overall Officials: marie migaud, PHD, Principal Investigator — University of South Alabama
Locations (1):
- University of South Alabama, Mobile, Alabama, United States

IPD SHARING:
Plan to Share IPD: No